CLINICAL TRIAL: NCT05595564
Title: Influence of Photobiomodulation on Anaerobic Capacity Under Normoxia and Hypoxia Conditions in Treadmill Runners
Brief Title: Influence of PBM on Anaerobic Capacity Under Normoxia and Hypoxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Hypoxia_PBM
Record Dates: First submitted 2022-10-18; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Low Level Laser Therapy; Photobiomodulation; Performance; Sport
Keywords: Physical Therapy; Photobiomodulation; Athletic Performance; Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoxia (Experimental): Participant developed running activity on a treadmill in hypoxic condition, submitted or not to photobiomodulation therapy.
  Interventions: Device: Photobiomodulation therapy
- Normoxia (Active Comparator): Participant developed treadmill running activity in normoxic condition, submitted or not to photobiomodulation therapy.
  Interventions: Device: Photobiomodulation therapy

INTERVENTIONS:
Device: Photobiomodulation therapy — A previous application of photobiomodulation therapy was offered or not, for possible performance enhancement.

SUMMARY:
The photobiomodulation (PBM) shows positive results in muscle performance, fatigue reduction, management of blood lactate production, analgesia and in the increase of VO2 maximal, favoring the increase of ATP production and thus the energy metabolism. The association of PBM applied before high-intensity treadmill training shows physiological improvements both in normoxic (Nor) and hypoxic (Hip) conditions. Anaerobic capacity (AC) is the maximum amount of ATP that can be resynthesized by anaerobic metabolism and is an important predictor of high-intensity exercise since an athlete's ability to perform efforts to increase maximal oxygen consumption (VO2max) depends on AL. In view of the above information the main objective of the present research project will be to investigate the effects of PBM on AC under normoxic and hypoxic conditions in amateur runners. To test the effects of exercise training on anaerobic capacity under normoxic and hypoxic conditions, 7 individuals will be randomly submitted to four maximal efforts to exhaustion with intensity corresponding to 110% of VO2max in Hip, Nor, Hip+Ebio and Nor+Ebio conditions. These efforts will be used to estimate the AC, that is, the maximum accumulated deficit of alternative oxygen (MAODRED), from the sum of the energy contribution of the anaerobic and lactic metabolisms.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* VO2 maximal equal to or greater than 34 ml/kg.min
* capacity for physical activity according to the PAR-Q questionnaire

Exclusion Criteria:

* musculoskeletal injury in the last three months;
* cardiovascular diseases;
* use of anabolic, anti-inflammatory and analgesic drugs 72 hours before the evaluations;
* use of alcohol and illicit drugs during the collection period;

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of excess oxygen consumption observed after exercise and blood lactate | 1 year
  To investigate the effects of photobiomodulation on anaerobic capacity in normoxia and hypoxia conditions in amateur runners

SECONDARY OUTCOMES:
Analysis of V02 max by a single supramaximal effort performed to exhaustion | 1 year
  To determine the alactic and lactic anaerobic and lactic anaerobic participation during exhaustive effort performed at 120% of VO2max in normoxia, hypoxia and with intervention of photobiomodulation

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Girasol, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The data will be shared in the form of the manuscript.

REFERENCES:
- [Background] Ferraresi C, Beltrame T, Fabrizzi F, do Nascimento ES, Karsten M, Francisco Cde O, Borghi-Silva A, Catai AM, Cardoso DR, Ferreira AG, Hamblin MR, Bagnato VS, Parizotto NA. Muscular pre-conditioning using light-emitting diode therapy (LEDT) for high-intensity exercise: a randomized double-blind placebo-controlled trial with a single elite runner. Physiother Theory Pract. 2015 Jul;31(5):354-61. doi: 10.3109/09593985.2014.1003118. Epub 2015 Jan 14. PMID 25585514
- [Background] Ando S, Komiyama T, Sudo M, Higaki Y, Ishida K, Costello JT, Katayama K. The interactive effects of acute exercise and hypoxia on cognitive performance: A narrative review. Scand J Med Sci Sports. 2020 Mar;30(3):384-398. doi: 10.1111/sms.13573. Epub 2019 Oct 27. PMID 31605635